CLINICAL TRIAL: NCT03867526
Title: Induced Pluripotent Stem Cells for the Development of Novel Drug Therapies for Hepatic and Neurological Wilson Disease
Brief Title: Establishment of Human Cellular Disease Models for Wilson Disease
Acronym: IPSWILSON
Status: Completed | Type: Observational
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: IPSWilson 06-2018
Record Dates: First submitted 2019-03-06; First posted 2019-03-08 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2020-04

CONDITIONS: Wilson Disease
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The skin biopsy will be carried out for patients with a diagnosis of Niemann Pick. The biopsy is performed by the physician by means of punch biopsy (diameter 2-3 mm) under local anesthesia, preferably on the forearm (alternatively: thigh). The biopsy is immediately transferred to sterile cell culture medium and sent by center representative for the quickest possible processing to CENTOGENE's laboratory located in Germany or to professional collaborators being part of the project.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Establishment of human cellular disease models for Wilson disease for an individualized therapy develop-ment having the capacity to address both hepatic and neurologic forms of the disease

DETAILED DESCRIPTION:
Wilson disease (WD) is caused by a defective gene for a copper-transporting protein that regulates cellular copper homeostasis in all major organs. Copper is an essential metal ion that is required for physiological cell functions (e.g. numerous enzymes require copper as a co-factor). It often occurs in people without a known family history of the condition.

The condition affects females and males likewise. Wilson disease occurs in approximately 1 out of every 30,000 births and belongs to the class of rare diseases. Because this is an inherited disorder, risks include a family history of Wilson disease.

Symptoms most often appear during adolescence or early adulthood. Symptoms may include:

increased thickness of the interventricular septum and left ventricular posterior wall supraventricular tachycardias tremors in hands, legs, head repetitive muscle contractions (dystonia) renal stones renal failure psychiatric symptoms (e.g. depression) liver disease

Therapeutic approaches include the drug Penicillamine, which binds to accumulated copper and eliminate it through urine. However, its use is controversy, since it is associated with an extended range of adverse effects and patients with neurologic manifestations deteriorated throughout the use of Penicillamine. Another strategy is the use of zinc salts that function via a detoxification effect of the stored copper ions. Recent studies suggested that zinc salts are effective in presymptomatic Wilson disease, but are problematic in hepatic Wilson disease and not suitable as a monotherapy.

In Wilson disease, the mutations of the hepatic copper transport ATP7B lead to a defective accumulation of copper in the cells. In addition to this primary pathological process, certain allelic variants (mutations in the protein-coding DNA region) are associated with the formation of a protein folding defect, often associated with considerable endoplasmic reticulum (ER) stress, which exposes the cell to a stress that leads to inflammatory reactions and in the worst case can lead to apoptotic cell death with the consequence of functional organ confinement, devastating disorders of whole organ systems and formation of tumors. Thus, ER stress can be involved in a substantial part of the clinical picture of the disease and support the progressive character of the disease. ER stress-associated protein mutants are generally able to re-spond to certain low-molecular-weight substances affecting cellular proteostasis. i.e. that the malignant influence of the misfolded protein on cellular physiology is mitigated or corrected.

A newly developed molecular therapeutic approach involves Pharmacological Chaperone therapy suitable to overcome protein misfolding and ER stress. The concept is that active-site binding low molecular competitive inhibitors (Pharmacological Chaperones) are able to stabilize the misfolded protein, bypass early degradation pathways (such as the ubiquitin-proteasome-system) and enhance/re-establish protein function at the site of action within the cell. These drugs are typically orally available, can reach even difficult to target organs (e.g. central nervous system) and are able to correct the pathophysiology. In addition to this class of inhibitory Pharmacological Chaperones, non-inhibitory PCs are being developed, because the multi-functional ATP7B protein provides distinct sites for a putative ligand binding.

A second class of low-molecular-weight substances target other components of the proteostasis network, e.g. the heat shock proteins or the proteasome as mediators to handle abnormally accumulated proteins within the ER.

Among the amenable protein folding diseases, the investigators investigated a few lysosomal storage dis-eases like Fabry, Gaucher and Pompe disease within recent years. A proof-of-concept study revealed Wilson disease as another pathology that can be addressed via this molecular therapeutic approach.

Therefore it is the goal of the study to prepare a cell culture from patients affected with Wil-son´s disease in order to identify novel pathways and proteins involved in disease progression that allow for an earlier diagnosis (i.e. before symptom onset) and that are suitable targets for an individualized therapeutic approach able to address not only the hepatic form, but also the neurologic form of the disease, which is less responsive to the current therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent will be obtained from the patient or the parents before any study related procedures.
* Patients of both genders older than 6 months and younger than 80 years
* The patient has a diagnosis of Wilson dis-ease

Exclusion Criteria:

* No Informed consent from the patient or the parents before any study related procedures
* Patients of both genders younger than 6 months and older than 80 years
* No diagnosis of Wilson disease

Ages: 6 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients has a diagnosis of Wilson disease
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Reprogramming patient-derived fibroblasts into induced pluripotent stem cells (iPSCs) | 12 months
  Generation of patient-specific iPSCs by using sendai-virus reprogramming method

SECONDARY OUTCOMES:
Differentiation of patient-specific iPSCs into disease-affected cell types | 24 months
  Establishment of iPSC-based disease model to recapitulate/phenocopy the disease in a dish

CONTACTS AND LOCATIONS:
Overall Officials: Arndt Rolfs, Prof. Dr., Principal Investigator — CENTOGENE GmbH Rostock
Locations (1):
- Childrens Hospital and Institute of Child Health, Ferozepur Road, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided